CLINICAL TRIAL: NCT02581956
Title: Walking Affecting Immunology and Quality of Life of Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Ming-Hsin Yeh, Attending Physician, Kaohsiung Veterans General Hospital.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS96-CT4-17
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: Immunology
MeSH Terms: conditions — Breast Neoplasms

ARMS (2):
- Walking Exercise (Experimental): For the exercise group, subjects were asked to follow a simple walking regimen. Walk normally with stable and comfortable stride rates during their exercise. The duration and frequency was initiated at a 30-minute or more daily exercise at least five days per week and gradually increased to a maximum of 60 minutes within subject's comfort zone.
  Interventions: Behavioral: Walking exercise
- No Intervention (Placebo Comparator): No exercise required
  Interventions: Behavioral: No walking exercise

INTERVENTIONS:
Behavioral: Walking exercise — Walk normally with the duration and frequency at a 30- minute or more daily at least five days per week and gradually increased to a maximum of 60 minutes daily.
  Arms: Walking Exercise
Behavioral: No walking exercise — no exercise
  Arms: No Intervention

SUMMARY:
Breast cancer is the leading cancer in women worldwide. The incidence of breast cancer is increasing probably due to the prolonged life expectancy and a variety of environmental factors. Fortunately, breast cancer outcome and survival are improving due to early detection and new treatment modalities. After making first strides against breast cancer, i.e. undergoing ablation surgery, most breast cancer survivors still have to go through a series of chemotherapy, which could prolong their survival but almost inevitably downgrade their quality of life due to grueling side effects, such as lack of energy and vulnerability to infection. Numerous medical interventions have been tried by healthcare providers to alleviate these side effects, but some of them are expensive and therefore become another burden for the cancer-afflicted patients. Previous studies have already indicated that exercise generated long-term benefits to breast cancer survivors, including improved physical functions, elevated maximal oxygen intake, decreases in lethargic symptom, increase in both immune function and quality of life. Among a variety of exercises, walking is the least costly, easy-to-follow type. Through a simple, predesigned walking regimen, the investigators expected that the breast cancer patients undergoing chemotherapy could cost-effectively reap some benefit either physically or psychologically.

Cluster of differentiation 3 (CD3+), presenting at all stages of T-cell development, is a useful maker to identify T-cells. (Cluster of differentiation 4)CD4+ T cells, also known as T helper cells, play an assistant role in the immunologic process, such as maturation of B cells, activations of macrophages or cytotoxic T cells. Cluster of differentiation 8 (CD8+) T cells, known as cytotoxic T cells, responsible for destroying virus-infected cells and tumor cells. Generally, the counts of CD3+ T cells, CD4+ T cells and CD8+ T cells could be a reflection of immune system health. Short-Form 36(SF-36), a patient-reported survey, is a widely adopted tool to evaluate patient's individual health status. By means of serial blood sample collections and the delivery of SF-36 survey, this study aimed to objectively and quantitatively evaluate the effects of aerobic walking on the breast cancer patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Stage I-II breast cancer
2. Have undergone ablative surgery
3. Going to receive chemotherapy

Exclusion Criteria:

* Difficulty walking

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
CD3, CD4, CD8 counts | through study completion, an average of 6 months
  CD3, CD4, CD8 counts during the chemotherapy periods
Quality of life measured by short-form36 | through study completion, an average of 6 months
  Quality of life measured by short-form 36